CLINICAL TRIAL: NCT01518088
Title: Effects of a Dietary Fiber on Human Gut Microbiota, Bioactive Metabolites and Blood Glucose Control
Brief Title: Effects of a Dietary Fiber on Fecal Microbiota and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PRT002
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2012-01

CONDITIONS: Focus of the Study is on Gut Health
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose dietary fiber (Experimental)
  Interventions: Dietary Supplement: Dietary Fiber
- High dose dietary fiber (Experimental)
  Interventions: Dietary Supplement: Dietary Fiber
- No added fiber (Placebo Comparator)
  Interventions: Dietary Supplement: Dietary Fiber

INTERVENTIONS:
Dietary Supplement: Dietary Fiber — Dietary fiber will be added to study foods

SUMMARY:
The purpose of the study is to examine how a dietary fiber affects metabolism in healthy overweight and obese adults. The fiber will be added to foods that participants will consume for two, three-week periods. The fiber will be given in two doses -- 15 g per day during one period, and 30 g per day in the other. In another three-week period, they will consume the same foods, but with no fiber added. Major outcomes will include fermentability of the fiber, as assessed by measurement of breath hydrogen, as well as shifts in fecal bacteria. The caloric value of the fiber will be determined and metabolic measures related to blood glucose control and inflammation will also be taken.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 25 to 35 kg/m2.
* Willing to consume study foods and comply with dietary exclusions and specimen collection

Exclusion Criteria:

* Pregnancy
* Diabetes
* Gastrointestinal disease
* Regular use of pre- or probiotics
* Recent use of antibiotics
* High intake of dietary fiber

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Metabolizable energy | 7 days, 3 times
  Urine and feces will be collected for 7 days at the end of each treatment period to allow for assessment of metabolizable energy
Fermentability | One, eight-hr day, three times
  Breath hydrogen will be measured hourly, over eight hours at the end of each treatment period

SECONDARY OUTCOMES:
Fecal microbiota | 2 days, three times, and 7 days, three times
  Fecal samples will be collected for 7 days at the end of each treatment period and for two days during washout periods
Blood glucose | For eight hours, three times
  An indwelling catheter will be placed and blood samples will be drawn over the course of an eight-hour period, at the end of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Keim, PhD, Principal Investigator — ARS/USDA, University of California - Davis
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States